CLINICAL TRIAL: NCT01716780
Title: Towards a Pain Free Hospital: Effect and Cost Effectiveness of Routine Screening and Treatment for Pain in Head and Neck Oncology Outpatients
Brief Title: Pain: Screen and Treat
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, RMH R&D, Dr John Williams, Royal Marsden NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR3439
Record Dates: First submitted 2012-09-12; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Head and Neck Cancer; Pain
MeSH Terms: conditions — Head and Neck Neoplasms; Pain | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine care (No Intervention): Patients allocated to the "control group" will undergo their 'usual care'; they will be given pain medication when they specifically request it or when their oncology doctor/ nurse or GP considers it appropriate to prescribe it, either at the oncology clinic visit or at any time during the course of the study.
- Intervention (Experimental): Patients allocated to the "intervention group" will be reviewed by the pain/palliative care team and will undergo prospective, proactive, integrated, structured pain treatment according to recent guidelines on cancer pain care.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Patients allocated to the "intervention group" will undergo prospective, proactive, integrated, structured pain treatment according to recent guidelines on cancer pain care
  Arms: Intervention

SUMMARY:
This study is looking at treating cancer pain in head and neck cancer. Patients are asked in outpatients to score their worst pain on a scale of 0 to 10 in the last 24 hours. Those with a pain score of 4 and above are randomised into the study.

Patients are allocated to continue with their current care (control group) or to be reviewed by the pain/palliative care team (intervention group). At baseline questionnaires are completed on level of pain, type of pain, quality of life and anxiety/depression. Information is also collected on the analgesia they've used in the past month and basic health economics (GP/hospital visits related to pain management and treatment).

Follow up in the trial is for 3 months and consists of questionnaires as above and further collection of information on analgesic usage and health economics.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending head and neck oncology clinics
* Patients with a cancer diagnosis who are receiving anti cancer treatment or who have received anti cancer treatment
* Patients who score 4 or more on the Brief Pain Inventory numerical rating scale screening question 'worst pain in past 24 hours'

Exclusion Criteria:

* age below 18 years
* patients unable to respond to an English written assessment
* patients with medical conditions that could affect their mental function or level of consciousness such as stroke, or dementia
* patients who score <4 on the Brief Pain Inventory numerical rating scale screening question
* patients already under the care of a pain/palliative care service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The change in pain score summarized from patient reports | 1 month, 2 months and 3 months

SECONDARY OUTCOMES:
Impact of pain | 1 month, 2 months, 3 months
  Measured by the brief pain inventory questionnaire
Adequacy of pain treatment | 1 month, 2 months and 3 months
  Using Pain Management Index, calculated from BPI and WHO ladder
Quality of life | 1 month, 2 months and 3 months
  Assessed using the EQ-5D questionnaire
Patient satisfaction | 1 month, 2 months and 3 months
  Likert scale
Anxiety and depression | 1 month, 2 months and 3 months
  Assessed using the Hospital anxiety and depression questionnaire
Treatment costs | 1 month, 2 months and 3 months
  Information collected on analgesic usage and contact with healthcare professionals for pain management purposes

CONTACTS AND LOCATIONS:
Overall Officials: John E Williams, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, London, United Kingdom